CLINICAL TRIAL: NCT02003690
Title: Dialectical Behavior Therapy (DBT) for Adolescents With Bipolar Disorder
Acronym: DBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tina R Goldstein, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH100056
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Dialectical Behavior Therapy + Pharmacotherapy; Standard of Care Psychotherapy + Pharmacotherapy
Keywords: Bipolar disorder; Adolescent suicidal behavior; Psychotherapy
MeSH Terms: conditions — Bipolar Disorder | interventions — Dialectical Behavior Therapy; Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical Behavior Therapy + Pharmacotherapy (Experimental): Dialectical Behavior Therapy + Pharmacotherapy
  Interventions: Behavioral: Dialectical Behavior Therapy; Other: Pharmacotherapy
- Standard of Care Psychotherapy + Pharmacotherapy (Active Comparator): Standard of Care Psychotherapy + Pharmacotherapy
  Interventions: Behavioral: Standard of Care Psychotherapy; Other: Pharmacotherapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Dialectical Behavior Therapy
  Arms: Dialectical Behavior Therapy + Pharmacotherapy
Behavioral: Standard of Care Psychotherapy — Standard of Care Psychotherapy
  Arms: Standard of Care Psychotherapy + Pharmacotherapy
Other: Pharmacotherapy — Standard of Care Pharmacotherapy

SUMMARY:
Of all psychiatric diagnoses, bipolar disorder imparts the greatest risk for completed suicide in adolescence, and is further associated with poor psychosocial functioning, substance abuse and legal difficulties, and exorbitant healthcare costs exceeding those for other adolescent psychiatric conditions. Treatment guidelines indicate optimal management of pediatric bipolar disorder includes a combination of medication and psychotherapy. Yet, little is known about effective psychotherapy approaches for this population, and none expressly target suicidality. An efficacious, cost-effective psychosocial intervention for adolescents with bipolar disorder has great potential to decrease the substantial morbidity, mortality and costs associated with adolescent bipolar disorder.

DETAILED DESCRIPTION:
Of all psychiatric diagnoses, bipolar disorder (BP) imparts the greatest risk for completed suicide in adolescence, and is associated with other negative outcomes including poor psychosocial functioning and substance abuse. Furthermore, healthcare costs for adolescents with BP exceed those for other adolescent psychiatric conditions. Treatment guidelines indicate optimal management of pediatric BP includes a combination of pharmacotherapy and psychotherapy. Yet, little is known about effective psychotherapy approaches for this population, and none expressly target suicidality. An efficacious, cost-effective psychotherapy for adolescents with BP has great potential to decrease the substantial morbidity, mortality and costs associated with this illness. Dialectical Behavior Therapy (DBT) is a skills-based psychotherapy originally developed for adults with borderline personality disorder. DBT holds promise for adolescents with BP given shared treatment targets including suicidality and psychosocial functioning. Our group's preliminary data on DBT for adolescents with BP provide strong support for the feasibility and acceptability of the treatment model, and indicate DBT is associated with improvement in targeted treatment domains including suicidality, emotional dysregulation, and depression, and these improvements are greater among adolescents receiving DBT as compared with standard of care (SOC) psychotherapy delivered at our Child and Adolescent Bipolar Services (CABS) specialty clinic. The proposed study aims to evaluate in a randomized controlled trial the efficacy of DBT + pharmacotherapy as compared with CABS SOC psychotherapy + pharmacotherapy over 2 year followup among adolescents (age 12-18) with BP (n=100). Primary outcome domains include suicidal events and mood symptoms. Our team includes an expert in health services cost effectiveness, enabling us to examine the cost effectiveness of DBT. Our exploratory aim is to elucidate moderators and mediators of DBT treatment response in this population. Identification of patient factors that predict response to DBT, as well as mechanisms by which DBT benefits patients, will directly inform the planful dissemination of the treatment (if shown to be effective) for those most likely to benefit. Furthermore, a supplement is enabling examination of neural mechanisms underlying DBT treatment response as assessed via fMRI at pre- and mid-treatment. These aims are in direct accord with the NIMH Strategic Plan to prioritize research on improved treatments for mental illness while also generating information regarding underlying mechanisms of disorder; facilitate widespread use of evidencebased interventions by demonstrating cost effectiveness; and systematically study elements of personalized intervention. Furthermore, this project aligns with the mission of the National Action Alliance for Suicide Prevention Research Prioritization Task Force: to prioritize gaps in the research that will reduce the rate of suicide and suicide attempts, to target particularly high-risk groups, and to move toward uptake of evidence-based interventions for suicidality.

ELIGIBILITY:
Inclusion Criteria: For the proposed study, inclusion criteria are as follows: 1) age 12 years, 0 months to 18 years, 11 months; 2) a diagnosis of Bipolar Disorder (BP) I, II or NOS by the K-SADS-PL with an acute manic, mixed or depressive episode in the 3 months preceding study entry; 3) willing to engage in pharmacotherapy treatment at the CABS specialty clinic; 4) at least one parent or guardian with whom the patient lives or interacts on a significant basis (5 hours per week or more) who is willing to participate in DBT skills training; 5) English language fluency and at minimum a 3rd grade literacy level; 6) able and willing to give informed consent/assent to participate.

Exclusion Criteria: For the proposed study, exclusion criteria are as follows: 1) evidence of mental retardation, pervasive developmental disorder, or organic central nervous system disorder by the K-SADS-PL, parent report, medical history, or school records; 2) a life-threatening medical condition requiring immediate treatment; 3) current victim of sexual or physical abuse.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Suicidal events | Over two year follow-up
  Suicidal events as assessed using the C-SSRS
Mood symptoms | Over two year follow-up
  As assessed using the KSADS-MRS and KSADS-DEP-P

SECONDARY OUTCOMES:
Cost effectiveness | Over two year follow-up
  Cost effectiveness as assessed using utilization and costs from the healthcare payer and provider system perspectives

CONTACTS AND LOCATIONS:
Overall Officials: Tina R Goldstein, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic / University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Goldstein TR, Axelson DA, Birmaher B, Brent DA. Dialectical behavior therapy for adolescents with bipolar disorder: a 1-year open trial. J Am Acad Child Adolesc Psychiatry. 2007 Jul;46(7):820-30. doi: 10.1097/chi.0b013e31805c1613. PMID 17581446
- [Derived] Goldstein TR, Merranko J, Rode N, Sylvester R, Hotkowski N, Fersch-Podrat R, Hafeman DM, Diler R, Sakolsky D, Franzen P, Birmaher B. Dialectical Behavior Therapy for Adolescents With Bipolar Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Jan 1;81(1):15-24. doi: 10.1001/jamapsychiatry.2023.3399. PMID 37703037